CLINICAL TRIAL: NCT02693132
Title: Comparison of Supervised and Unsupervised Physical Activity Programs During a Standard Behavioral Weight Loss Intervention for Adults Who Are Overweight or Obese
Brief Title: Comparison of Supervised and Unsupervised Physical Activity Programs During a Weight Loss Intervention for Adults
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO15110570
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Obesity
Keywords: Obesity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supervised (SUP-PA) (Experimental): Weight loss intervention that focuses on supervised physical activity and involves an energy restricted diet. Physical activity will be supervised by trained staff.
  Interventions: Behavioral: Supervised (SUP-PA)
- Unsupervised (UNSUP-PA) (Experimental): Weight loss intervention that focuses on unsupervised physical activity (identical dose to SUP-PA) and involves an energy restricted diet (identical diet to SUP-PA). Physical activity will be self-monitored but no activity tracker will be used as an intervention tool.
  Interventions: Behavioral: Unsupervised (UNSUP-PA)
- Step-based (STEP) (Experimental): Weight loss intervention that focuses on unsupervised physical activity prescribed as steps/day and involves an energy restricted diet (identical diet to SUP-PA and UNSUP-PA). Physical activity will be self-monitored and a pedometer will be used to track steps/day.
  Interventions: Behavioral: Step-based (STEP)

INTERVENTIONS:
Behavioral: Supervised (SUP-PA) — Weight loss intervention that involves an energy restricted diet plus the inclusion of 150 minutes per week of supervised moderate-to-vigorous intensity physical activity.
  Arms: Supervised (SUP-PA)
Behavioral: Unsupervised (UNSUP-PA) — Weight loss intervention that involves an energy restricted diet plus the inclusion of 150 minutes per week of unsupervised moderate-to-vigorous intensity physical activity.
  Arms: Unsupervised (UNSUP-PA)
Behavioral: Step-based (STEP) — Weight loss intervention that involves an energy restricted diet plus the inclusion of physical activity in the form of 10,000 steps/day with 2,500 "brisk" steps/day.
  Arms: Step-based (STEP)

SUMMARY:
Adults who are overweight or obese are typically prescribed a calorie-restricted diet and physical activity to promote weight loss and improve health. The manner in which physical activity is prescribed and monitored may influence physical activity engagement. Within the context of clinical research, physical activity has been prescribed in either a supervised or unsupervised manner. Supervised physical activity is typically done in a health-fitness facility under the direct supervision of trained staff. The alternative, unsupervised physical activity, promotes physical activity participation in a setting that is convenient to the individual. Unsupervised activity can be done in any environment or at any time that best suits the individual. Knowing the effects of unsupervised physical activity is important because of the translation of this type of physical activity to non-research settings. Therefore, knowing the magnitude of the physiological effects of unsupervised physical activity compared to supervised physical activity at the same prescribed intensity and dose is of clinical and public health importance. This study is designed to provide insight on these important research questions that can inform future research and the application to clinical, public health, and health-fitness settings.

DETAILED DESCRIPTION:
Approximately 69% of the U.S. adult population is overweight, defined by a body mass index (BMI) of ≥ 25.0 kg/m2, and 35% are obese (BMI ≥ 30.0 kg/m2), with the prevalence of overweight and obesity rising drastically over the past several decades. Adults who are overweight or obese are typically recommended to change lifestyle factors (e.g. diet, physical activity, etc.) to lose weight and improve health. When evaluating the effects of these lifestyle changes on weight and health in a research setting, physical activity is supervised (i.e. physical activity completed in a health-fitness facility with direct supervision from trained staff). With supervised physical activity, researchers are able to quantify the frequency, intensity, duration, and type of physical activity. Thus, supervised physical activity is considered the gold-standard when evaluating the effects of physical activity on weight and other physiological parameters. However, the results of supervised physical activity trials may not translate to clinical settings. A typical clinical approach prescribes physical activity in an unsupervised manner (i.e. physician tells patient to be more physically active or take more steps/day). Unsupervised physical activity can be done in any environment or at any time that best suits the individual. Knowing the effects of unsupervised physical activity is important because of the translation of this type of physical activity to non-research settings. Therefore, knowing the magnitude of the physiological effects of unsupervised physical activity compared to supervised physical activity at the same prescribed intensity and dose is of clinical and public health importance especially in an overweight and obese population. This study is designed to provide insight on these important research questions that can inform future research and the application to clinical, public health, and health-fitness settings.

Participants will be randomized to one of three groups: supervised physical activity prescribed in min/week (SUP-PA), unsupervised physical activity prescribed in min/week (UNSUP-PA), and unsupervised physical activity prescribed in steps/day (STEP). Participants in all three groups will participate in a behavioral weight loss intervention which includes dietary counseling and weekly group sessions during the 12-week program. SUP-PA will be prescribed 150 minutes/week of moderate-to-vigorous physical activity (MVPA) completed under direct supervision of trained staff at a designated health-fitness facility. UNSUP-PA will be prescribed a physical activity dose matched to SUP-PA. STEP will be prescribed a 10,000 step/day recommendation with 2,500 of those steps completed at a "brisk" pace. The primary aim of this study is to compare the effects of all three groups on moderate-to-vigorous physical activity (MVPA) accumulated in bouts of at least 10 minutes. The primary outcome will be assessed at baseline, week 4, week 8, and week 12. Secondary aims of this trial include comparing light intensity physical activity, sedentary time, cardiorespiratory fitness, weight, body composition, waist circumference measures, physical activity self-efficacy, blood pressure, and dietary intake across all three groups. Secondary aims will be assessed at baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 18-55 years old
* BMI of 25.0 to <40.0 kg/m2
* Ability to provide informed consent
* Ability to provide physician's clearance to participate in a weight loss intervention

Exclusion Criteria:

* Engaging in >60 min/wk (accumulated in bouts of ≥10 minutes) of moderate-to-vigorous physical activity over the past month
* Presence of contraindications to physical activity as identified on a physical activity readiness questionnaire (PAR-Q)
* History of metabolic, cardiac, or pulmonary disease that classifies the individual as high risk by the American College of Sports Medicine (e.g., coronary heart disease, diabetes mellitus, uncontrolled hypertension, etc.)
* History of myocardial infarction, coronary bypass surgery, angioplasty, or other cardiovascular- related surgeries.
* Taking medication that may affect heart rate or blood pressure responses to physical activity
* Resting systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg.
* Medication that may affect body weight/metabolism (e.g., synthroid).
* Current or previous participation in a physical activity or weight management research project in the past 6 months
* Weight loss of ≥5% or 15 pounds total of current body weight in the previous 6 months.
* Currently being treated for an eating disorder (e.g., anorexia, bulimia, etc.)
* Previously undergone bariatric surgery (e.g., lap-band, gastric bypass, etc.)
* For women, those currently pregnant, pregnant during the previous 6 months, or plan on becoming pregnant in the next 6 months
* Currently being treated for any psychological issues or problems, taking any psychotropic medications, or receiving treatment with psychotropic medications within the previous 6 months.
* Being out of town during for an extended amount of time during the weight loss intervention which may affect participation in the study
* Currently using a physical activity monitor to track activity (e.g., Jawbone UP, Fitbit, etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Creasy, Principal Investigator — University of Pittsburgh; John M Jakicic, Study Chair — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Started | 17 | 17 | 18
Completed | 16 | 16 | 17
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP) | Total
Number analyzed (Participants) | 17 | 17 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (8.5) | 46.2 (10.1) | 39.3 (10.7) | 43.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 13 | 38
  Male | 4 | 5 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 3 | 12
  White | 12 | 11 | 12 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate-to-Vigorous Physical Activity (Accumulated in Bouts of at Least 10 Minutes)
Description: Measured using a wearable device and by questionnaire
Time Frame: Baseline (0 weeks), 4 Weeks, 8 Weeks, 12 Weeks
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Number analyzed (Participants) | 16 | 16 | 17
minutes/day
  Baseline | 28.0 (23.5) | 25.6 (36.0) | 35.4 (33.5)
  4 Weeks | 44.4 (24.0) | 38.3 (42.6) | 42.8 (23.6)
  8 Weeks | 54.3 (37.2) | 46.1 (45.5) | 51.2 (33.5)
  12 Weeks | 49.6 (38.7) | 41.7 (44.5) | 47.0 (28.2)
Statistical Analysis 1: Comparison: Supervised (SUP-PA) vs Unsupervised (UNSUP-PA) vs Step-based (STEP); Test type: Superiority; p < 0.05, ANOVA

2. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Measured using a submaximal graded exercise test on a treadmill, with termination occurring at 85% of age-predicted maximal heart rate (computed at [220-age]*0.85]). The outcome was measures as oxygen consumption (ml/kg/min) at the point of test termination.
Time Frame: Baseline (0 weeks),12 Weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Number analyzed (Participants) | 16 | 16 | 17
ml/kg/min
  Baseline | 24.4 (4.2) | 23.9 (4.5) | 27.9 (5.5)
  12 Weeks | 28.2 (4.9) | 27.7 (5.7) | 29.2 (6.0)
Statistical Analysis 1: Comparison: Supervised (SUP-PA) vs Unsupervised (UNSUP-PA) vs Step-based (STEP); Test type: Superiority; p < 0.05, ANOVA

3. Secondary Outcome: Change in Body Weight
Description: Measured in kilograms using a digital scale
Time Frame: Baseline (0 weeks),12 Weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Number analyzed (Participants) | 16 | 16 | 17
kilograms
  Baseline | 84.0 (13.7) | 86.8 (13.1) | 87.7 (14.7)
  12 Weeks | 80.1 (13.2) | 81.6 (11.8) | 82.3 (14.1)
Statistical Analysis 1: Comparison: Supervised (SUP-PA) vs Unsupervised (UNSUP-PA) vs Step-based (STEP); Test type: Superiority; p < 0.05, ANOVA

4. Secondary Outcome: Change in Fat Mass
Description: Measured as fat mass (kg) using dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline (0 weeks),12 Weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Number analyzed (Participants) | 16 | 16 | 17
kilograms
  Baseline | 34.6 (6.7) | 35.4 (7.6) | 33.7 (6.3)
  12 Weeks | 30.8 (6.4) | 31.3 (8.2) | 29.6 (6.2)
Statistical Analysis 1: Comparison: Supervised (SUP-PA) vs Unsupervised (UNSUP-PA) vs Step-based (STEP); Test type: Superiority; p < 0.05, ANOVA

5. Secondary Outcome: Change in Energy Intake
Description: Measured as kcal/day using a questionnaire
Time Frame: Baseline (0 weeks),12 Weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
Number analyzed (Participants) | 14 | 16 | 17
kcal/day
  Baseline | 1774 (679) | 1773 (922) | 1885 (905)
  12 Weeks | 1214 (370) | 1342 (438) | 1497 (522)
Statistical Analysis 1: Comparison: Supervised (SUP-PA) vs Unsupervised (UNSUP-PA) vs Step-based (STEP); Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected during the 3 months of the intervention
Arm/Group | Supervised (SUP-PA) | Unsupervised (UNSUP-PA) | Step-based (STEP)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes